CLINICAL TRIAL: NCT05334342
Title: Two Birds with One Stone: Impact of a Low Glycemic Index Diet on Postprandial Hypotension and Glucose Metabolism in Individuals with Spinal Cord Injury
Brief Title: Low-GI Diet Vs High-GI Diet in Individuals with SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jia Li, Principle Investigator, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-300008930
Record Dates: First submitted 2022-03-21; First posted 2022-04-19 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Spinal Cord Injuries; Postprandial Hypotension; Glucose Metabolism Disorders
Keywords: Spinal Cord Injury; Low glycemic index diet
MeSH Terms: conditions — Spinal Cord Injuries; Glucose Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: The investigator(s) propose to recruit 12 participants with chronic SCI (>1 year) and utilize a single-blinded randomized crossover design (low-GI vs. high-GI diet) to assess postprandial BP and postprandial glycemic responses to the study diets in this population.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The random permuted blocks strategy will be used in this study to randomly allocate an equal number of participants into the two crossover arms by the study statistician. Diet group assignment will be coded (e.g., low-gi diet=diet a; high-gi diet=diet b). Only the kitchen staff preparing the meals will know the code. Study personnel analyzing the biological samples, entering data, and performing statistical analyses will be blinded to the diet group assignment to reduce bias. Due to the nature of dietary studies, participants will not be blinded to the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-GI Diet (Experimental): Low Glycemic Index Diet
  Interventions: Dietary Supplement: Low-GI Diet
- High-GI Diet (Active Comparator): High Glycemic Index Diet
  Interventions: Dietary Supplement: High-GI Diet

INTERVENTIONS:
Dietary Supplement: Low-GI Diet — Participants will be given a low glycemic index diet
  Arms: Low-GI Diet
Dietary Supplement: High-GI Diet — Participants will be given a high glycemic index diet
  Arms: High-GI Diet

SUMMARY:
The purpose of this pilot research project is to examine the impact of a low-glycemic index (GI) diet on postprandial hypotension and glucose control in individuals with chronic spinal cord injury. The objectives are: 1) To evaluate the effect of the low-GI diet on the magnitude of postprandial systolic blood pressure drop compared to a high-GI control diet. 2)To evaluate the effect of a low-GI diet on postprandial glucose and insulin responses compared to a high-GI control diet.

DETAILED DESCRIPTION:
Participants will first come for a screening visit one time, lasting a total of 2.5hours. For this screening visit, each participant will need to fast for 12 hours(go 12 hours without eating from the last meal). During this study visit, each participant will be going through the following tests:

* Urine pregnancy tests (for females)
* Medical History Questionnaire: It will take about 10 minutes, and participants will fill out a 1-page questionnaire about their medical history and medication use
* Each participant will consume a semi-liquid meal within 5 minutes
* Each participant's blood pressure will be measured every 5 minutes before eating, for 15 minutes, and for 2 hours after eating.

After the screening visit, each participant will be coming for study visits on 2 separate mornings, separated by at least 1 week. On these two mornings, the participant will be randomly picked (like the flip of a coin) by a computer to eat the low-glycemic index meal or high-glycemic index meal. After the visit in the morning, the participant will be sent home wearing a blood pressure monitor and blood sugar monitor, along with study meals the participant will be eating for 3 days.

These procedures and tests will be made during these 3-day periods:

At UAB during the morning visit:

* Meal tolerance test: Firstly, a nurse will place an intravenous catheter in the participant's arm to allow blood draws. The participant will be asked to eat the study meal given by the investigators, and provide several blood samples (immediately before and 10, 30, 60, 90, and 120 minutes after glucose ingestion). The total amount of blood taken will be about 3 tablespoons.
* Participant's blood pressure will be measured every 5 minutes before eating, for 15 minutes, and for 2 hours after eating.

After participant goes home from UAB:

* Before the participant leaves for home, the investigator(s) will fit a wearable blood pressure monitor on his/her arm and insert a continuous glucose monitor in the back of the other arm.
* The blood pressure monitors will be programmed to measure blood pressure every 15 minutes during the daytime and hourly during nighttime. The daytime and nighttime cycle will be set according to each participant's sleep/wake pattern. Participants will need to keep the monitored arm steady and at heart level during each blood pressure reading.
* Each participant will be provided with meals for 3 days. They will be eating all and only the meals the investigators provide during these 3 days.
* Each participant will be filling out a checklist to record the time of each meal consumed.
* Each participant will be asked questions regarding their daily activity for the past 3 days for the investigators to estimate their activity level. The investigators will use the Physical Activity Recall Assessment for People with Spinal Cord Injury (PARA-SCI) questionnaire. This takes about 30 minutes and will be done over the phone

ELIGIBILITY:
Inclusion Criteria:

* Chronic SCI, At least 1 year after injury, Injury level between Cervical 4 and Lumbar 2, with an American Spinal Injury Association (ASIA) Impairment Scale classification of A-D

Exclusion Criteria:

* pregnancy or breastfeeding, type 1 or insulin-dependent type 2 diabetes, a recent change in the use of any medications, previous diagnosis of heart diseases and/or stroke, or neurological impairment other than SCI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Post-meal Systolic Blood Pressure Change- Visit 1 | In-lab testing - Visit 1 - Day 1
  SBP will be measured in the temperature-controlled, quiet, dimly lit room. Measurements will be taken using an automated sphygmomanometer every 5 minutes for 20 minutes before, and for 120 minutes after meal intake, with the participant in a sitting position. Investigators will identify the nadir of SBP during the 120-minute postprandial period. The magnitude of the drop in SBP will be calculated by subtracting the nadir value from the resting baseline average value.
Post-meal Systolic Blood Pressure Change- Visit 2 | In-lab testing - Visit 2 - Day 1
  SBP will be measured in the temperature-controlled, quiet, dimly lit room. Measurements will be taken using an automated sphygmomanometer every 5 minutes for 20 minutes before, and for 120 minutes after meal intake, with the participant in a sitting position. Investigators will identify the nadir of SBP during the 120-minute postprandial period. The magnitude of the drop in SBP will be calculated by subtracting the nadir value from the resting baseline average value.
Low-GI Diet on Post-meal Systolic Blood Pressure Change- Diet A- Day 1 | Free-living condition - Diet A - Day 1
  After the in-lab meal test, each participant will be fitted with an ambulatory blood pressure (ABP) monitoring (ABPM) device, the Spacelabs OnTrak device, which has been validated for use in assessing ABP. The first measurement will be obtained at UAB to ensure proper function of the device. Each participant's ABP will be monitored for a total of 3 days. The monitors will be programmed to measure BP at 15-minute intervals during the daytime (while participants are awake, e.g., 6 am to 11 pm). Participants will be instructed to keep the monitored arm steady and at heart level during each BP reading. Investigators will utilize the menu checklist to identify the timing of each meal consumed. The magnitude of the PPH will be calculated for each meal, by substracting the nadir of SBP within 2 hours after each meal from the average SBP before each meal.
Low-GI Diet on Post-meal Systolic Blood Pressure Change- Diet A- Day 2 | Free-living condition - Diet A - Day 2
  After the in-lab meal test, each participant will be fitted with an ABPM device, the Spacelabs OnTrak device, which has been validated for use in assessing ABP. The first measurement will be obtained at UAB to ensure proper function of the device. The monitors will be programmed to measure BP at 15-minute intervals during the daytime (while participants are awake, e.g., 6 am to 11 pm). Participants will be instructed to keep the monitored arm steady and at heart level during each BP reading. Investigators will utilize the menu checklist to identify the timing of each meal consumed. The magnitude of the PPH will be calculated for each meal, by substracting the nadir of SBP within 2 hours after each meal from the average SBP before each meal.
Low-GI Diet on Post-meal Systolic Blood Pressure Change- Diet A- Day 3 | Free-living condition - Diet A - Day 3
  After the in-lab meal test, each participant will be fitted with an ABPM device, the Spacelabs OnTrak device, which has been validated for use in assessing ABP. The first measurement will be obtained at UAB to ensure proper function of the device. The monitors will be programmed to measure BP at 15-minute intervals during the daytime (while participants are awake, e.g., 6 am to 11 pm). Participants will be instructed to keep the monitored arm steady and at heart level during each BP reading. Investigators will utilize the menu checklist to identify the timing of each meal consumed. The magnitude of the PPH will be calculated for each meal, by substracting the nadir of SBP within 2 hours after each meal from the average SBP before each meal.
Low-GI Diet on Post-meal Systolic Blood Pressure Change- Diet B- Day 1 | Free-living condition - Diet B - Day 1
  After the in-lab meal test, each participant will be fitted with an ABPM device, the Spacelabs OnTrak device, which has been validated for use in assessing ABP. The first measurement will be obtained at UAB to ensure proper function of the device. The monitors will be programmed to measure BP at 15-minute intervals during the daytime (while participants are awake, e.g., 6 am to 11 pm). Participants will be instructed to keep the monitored arm steady and at heart level during each BP reading. Investigators will utilize the menu checklist to identify the timing of each meal consumed. The magnitude of the PPH will be calculated for each meal, by substracting the nadir of SBP within 2 hours after each meal from the average SBP before each meal.
Low-GI Diet on Post-meal Systolic Blood Pressure Change- Diet B- Day 2 | Free-living condition - Diet B - Day 2
  After the in-lab meal test, each participant will be fitted with an ABPM device, the Spacelabs OnTrak device, which has been validated for use in assessing ABP. The first measurement will be obtained at UAB to ensure proper function of the device. The monitors will be programmed to measure BP at 15-minute intervals during the daytime (while participants are awake, e.g., 6 am to 11 pm). Participants will be instructed to keep the monitored arm steady and at heart level during each BP reading. Investigators will utilize the menu checklist to identify the timing of each meal consumed. The magnitude of the PPH will be calculated for each meal, by substracting the nadir of SBP within 2 hours after each meal from the average SBP before each meal.
Low-GI Diet on Post-meal Systolic Blood Pressure Change- Diet B- Day 3 | Free-living condition - Diet B - Day 3
  After the in-lab meal test, each participant will be fitted with an ABPM device, the Spacelabs OnTrak device, which has been validated for use in assessing ABP. The first measurement will be obtained at UAB to ensure proper function of the device. The monitors will be programmed to measure BP at 15-minute intervals during the daytime (while participants are awake, e.g., 6 am to 11 pm). Participants will be instructed to keep the monitored arm steady and at heart level during each BP reading. Investigators will utilize the menu checklist to identify the timing of each meal consumed. The magnitude of the PPH will be calculated for each meal, by substracting the nadir of SBP within 2 hours after each meal from the average SBP before each meal.

SECONDARY OUTCOMES:
Low-GI diet on postprandial glycemia- Visit 1 | In-Lab testing - Visit 1 - Day 1
  The investigators will obtain blood samples to assess blood sugar and insulin responses to the study diet throughout the in-lab testing period. An intravenous catheter will be in an antecubital vein for blood draws 10 minutes before and 10, 30, 60, 90, and 120 minutes after meal consumption.
Low-GI diet on postprandial glycemia - Visit 2 | In-Lab testing - Visit 2 - Day 1
  The investigators will obtain blood samples to assess blood sugar and insulin responses to the study diet throughout the in-lab testing period. An intravenous catheter will be in an antecubital vein for blood draws 10 minutes before and 10, 30, 60, 90, and 120 minutes after meal consumption.
Low-GI Diet on Postprandial Glucose Responses | Free-living condition - Diet A - Day 2
  After the standard lab meal test, an FDA-approved CGM device (Dexcom G6 Pro, Dexcom, Inc.) will be placed in the back of each participant's arm to automatically measure glucose every 5 minutes during the 3-day study period. Postprandial peak glucose concentration and glucose area under the curve within 2 hours after each meal will be identified and calculated (mealtime will be recorded on the menu checklist by each participant or their caregiver).
Low-GI Diet on Postprandial Glucose Responses | Free-living condition - Diet A - Day 3
  After the standard lab meal test, an FDA-approved CGM device (Dexcom G6 Pro, Dexcom, Inc.) will be placed in the back of each participant's arm to automatically measure glucose every 5 minutes during the 3-day study period. Postprandial peak glucose concentration and glucose area under the curve within 2 hours after each meal will be identified and calculated (mealtime will be recorded on the menu checklist by each participant or their caregiver).
Low-GI Diet on Postprandial Glucose Responses | Free-living condition - Diet B - Day 2
  After the standard lab meal test, an FDA-approved CGM device (Dexcom G6 Pro, Dexcom, Inc.) will be placed in the back of each participant's arm to automatically measure glucose every 5 minutes during the 3-day study period. Postprandial peak glucose concentration and glucose area under the curve within 2 hours after each meal will be identified and calculated (mealtime will be recorded on the menu checklist by each participant or their caregiver).
Low-GI Diet on Postprandial Glucose Responses | Free-living condition - Diet B - Day 3
  After the standard lab meal test, an FDA-approved CGM device (Dexcom G6 Pro, Dexcom, Inc.) will be placed in the back of each participant's arm to automatically measure glucose every 5 minutes during the 3-day study period. Postprandial peak glucose concentration and glucose area under the curve within 2 hours after each meal will be identified and calculated (mealtime will be recorded on the menu checklist by each participant or their caregiver).

CONTACTS AND LOCATIONS:
Overall Officials: Jia Li, PhD, Principal Investigator — The University of Alabama at Birmingham Department of Physical Medicine and Rehabilitation
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers that are not on the study.